CLINICAL TRIAL: NCT03717922
Title: Low Intensity Focused Ultrasound of Medial Temporal Lobe Regions for the Improvement of Learning and Memory / Low Intensity Focused Ultrasound as a Non-Invasive Neural Prosthetic for the Improvement of Emotion Regulation
Brief Title: Low Intensity Focused Ultrasound for Learning and Memory and Emotion Regulation
Acronym: LIFUPMEMEMOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Taylor Kuhn, Adjunct Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB#18-000104 / IRB#18-000978; NCT03782194 (obsolete NCT alias)
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Brain Diseases; Memory Disorders; Learning Disabilities; Cognitive Impairment
Keywords: Ultrasound; MRI; Learning; Memory; Cognitive Neural Prosthetic
MeSH Terms: conditions — Brain Diseases; Memory Disorders; Learning Disabilities; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to both study arms; the order in which they complete the arms will be randomized and counterbalanced. The two visits will be spaced apart by 2 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to exactly when the transducer is turned on, and to the region being targeted at each visit. The individual collecting the neuropsychological data will be blinded to which condition (amygdala, entorhinal cortex) the participant completed during the session. The statistical analysts for both the neuropsychological and neuroimaging data will also be blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Amygdala first, then Entorhinal Cortex (Experimental): Low Intensity focused ultrasound pulsation (LIFUP) will be administered to the amygdala while participants are in the MRI scanner. Then, 2 weeks later, entorhinal cortex LIFUP will be administered.
  Interventions: Device: Low Intensity Focused Ultrasound Pulsation to Amygdala; Device: Low Intensity Focused Ultrasound Pulsation to Entorhinal Cortex
- Entorhinal Cortex first, then Amygdala (Experimental): Low Intensity focused ultrasound pulsation (LIFUP) will be administered to the entorhinal cortex while participants are in the MRI scanner. Then, 2 weeks later, amygdala LIFUP will be administered.
  Interventions: Device: Low Intensity Focused Ultrasound Pulsation to Amygdala; Device: Low Intensity Focused Ultrasound Pulsation to Entorhinal Cortex

INTERVENTIONS:
Device: Low Intensity Focused Ultrasound Pulsation to Amygdala — Low intensity focused ultrasound pulsation will be administered to the amygdala in 10 sonications at 650kHz, ispta 720mW/cm, pulse repetition frequency 10Hz, duty cycle 5% duration 30s, with 30s spacing between sonications. Prior to receiving LIFUP sonication, the LIFUP transducer will be aimed at the amygdala and gently strapped in place to their head. Participants will then return to the scanner where a T1 image will verify the position of the LIFUP transducer and allow for estimation of the spatial location of the sonication beam focus. If needed, adjustments to transducer placement will be made to ensure that the beam focus is correctly aimed; an additional T1 will be collected after adjustment. Once correct placement of the transducer has been confirmed, LIFUP will be administered.
Device: Low Intensity Focused Ultrasound Pulsation to Entorhinal Cortex — Low intensity focused ultrasound pulsation will be administered to the entorhinal cortex in 10 sonications at 650kHz, ispta 720mW/cm, pulse repetition frequency 100Hz, duty cycle 5% duration 30s, with 30s spacing between sonications. Prior to receiving LIFUP sonication, the LIFUP transducer will be aimed at the entorhinal cortex and gently strapped in place to their head. Participants will then return to the scanner where a T1 image will verify the position of the LIFUP transducer and allow for estimation of the spatial location of the sonication beam focus. If needed, adjustments to transducer placement will be made to ensure that the beam focus is correctly aimed; an additional T1 will be collected after adjustment. Once correct placement of the transducer has been confirmed, LIFUP will be administered.

SUMMARY:
The goal of this clinical trial is to investigate the impact of low intensity focused ultrasound pulsation (LIFUP) to two different brain regions, the amygdala and entorhinal cortex, in older adults. The main questions it aims to answer are:

1. Will LIFUP change brain activity in the targeted regions?
2. Will LIFUP to the amygdala have an impact on anxiety and emotion regulation?
3. Will LIFUP to the entorhinal cortex have an impact on memory performance?

Participants will complete two in-person visits including neuropsychological testing, MRI of the brain, and LIFUP to the brain.

DETAILED DESCRIPTION:
Medial temporal lobe (MTL)-dependent memory is impacted by a wide range of psychiatric and neurologic conditions. These cognitive limitations often result in limited functional abilities for patients. Currently available pharmacologic and behavioral treatments are somewhat controversial and have minimal evidence-based effectiveness. Recently, deep brain stimulation was used to modulate MTL activity and subsequently improve memory performance. However, such implantable devices require neurosurgery with major associated health risk. At present, there are no publications reporting non-invasive neurostimulation targeting MTL regions to improve memory. The central hypothesis of this project is that non-invasive, low intensity focused ultrasound pulsation (LIFUP) can selectively increase regional MTL activity and thus be used as a cognitive neural prosthetic capable of improving memory performance. The aims of this portion of the study focus on whether LIFUP can increase blood oxygen level dependent (BOLD) activation and perfusion (measured by arterial spin labeling) in the entorhinal cortex and functionally associated regions, and whether LIFUP to the entorhinal cortex will result in improved memory.

The Amygdala is highly involved in emotional response, emotional reactivity and anxiety. Amygdala functions are therefore involved in a wide range of psychiatric disorders including generalized and social anxiety, specific phobia, obsessive compulsive disorder and posttraumatic stress disorder. Therefore, potential clinical implications of amygdala stimulation are great. However, to date, such efforts have been limited by the inability of non-invasive neuromodulation techniques (e.g. transcranial magnetic stimulation - TMS) to reach the amygdala and the highly invasive (i.e. neurosurgical) nature of methods (e.g. deep brain stimulation - DBS) which can, but to our knowledge has rarely been used, target these areas. In order to overcome these current limitations, study investigators propose the use of low intensity focused ultrasound pulsation (LIFUP) to affect amygdala activity to improve emotion regulation. The aim of this portion of the study focuses on whether LIFUP can modulate blood oxygen level dependent (BOLD) activation and perfusion (measured by arterial spin labeling) in the amygdala and functionally associated regions, and whether LIFUP to the amygdala will result in changes to anxiety levels and emotion regulation.

This study will be conducted using a crossover design in which each participant will complete two visits spaced two weeks apart. At one visit, they will receive LIFUP sonication (with parameters hypothesized to be inhibitory) to the right amygdala, and at the other, they will receive sonication (with parameters hypothesized to be excitatory) to the left entorhinal cortex. The order of conditions will be randomized and counterbalanced across participants. Participants will be blinded to condition order, and all other testing will be conducted the same at both visits. This design will allow us to test the effects of two potentially clinically-relevant targets for LIFUP, and will allow us to determine whether observed effects on brain activity, learning and memory, and emotion regulation are target-specific by comparing results between the two LIFUP paradigms.

ELIGIBILITY:
Inclusion Criteria:

* Must be right handed
* English must be the dominant language

Exclusion Criteria:

* contraindications for MRI (e.g. metal implants, pregnancy)
* history of head injury sufficient to warrant medical attention
* history of alcohol abuse or dependence
* history of substance abuse or dependence
* history of major psychiatric illness requiring treatment
* history of cancer or other neoplastic syndromes
* history of major neurologic illness (e.g. epilepsy).

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taylor P Kuhn, PhD, Principal Investigator — UCLA Longevity Center
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amygdala First, Then Entorhinal Cortex | Entorhinal Cortex First, Then Amygdala
Started | 10 | 11
Completed Visit 1 | 10 | 11
Completed (Completed Visits 1 & 2) | 8 | 9
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amygdala First, Then Entorhinal Cortex | Entorhinal Cortex First, Then Amygdala | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (8.2) | 61.2 (9.5) | 60.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 6 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 3 | 8
  Black or African American | 2 | 1 | 3
  Asian | 1 | 1 | 2
  Hispanic or Latino | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Rey Auditory Verbal Learning Task
Description: The Rey Auditory Verbal Learning Task is an assessment of verbal memory in which a list of 15 words is presented 5 times and participants are asked to repeat all the words they can remember immediately after each list presentation. This is followed by presentation and recall of an interference list. Immediately after the interference trial, the participant is asked to recall the original list. Then, 20 minutes later, they are asked to recall the original list again (delayed recall).
  "Learning Trials Total": Total number of words learned / successfully recalled across the five learning trials plus the post-interference immediate recall trial. This score does not include the words recalled from the interference list.
  "Delayed Recall": Total number of words recalled during the delayed recall trial of the Rey Auditory Verbal Learning Task
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Population: All participants who completed this assessment before and after LIFUP at both the entorhinal cortex and the amygdala visits were included in analyses
Measure: Mean (Standard Deviation); unit: Words Recalled
Groups:
- LIFUP to Entorhinal Cortex: LIFUP will be administered to the entorhinal cortex in 10 sonications at 650kHz, 720mW/cm, duty cycle 5%, pulse repetition frequency 100Hz, duration 30s, with 30s spacing between sonications.
- LIFUP to Amygdala: LIFUP will be administered to the amygdala in 10 sonications at 650kHz, 720mW/cm, duty cycle 5%, pulse repetition frequency 10Hz, duration 30s, with 30s spacing between sonications.
Arm/Group | LIFUP to Entorhinal Cortex | LIFUP to Amygdala
Number analyzed (Participants) | 17 | 17
Words Recalled
  Pre-LIFUP Learning Trials Total | 50.00 (11.09) | 50.29 (9.79)
  Post-LIFUP Learning Trials Total | 47.59 (9.21) | 47.88 (11.10)
  Pre-LIFUP Delayed Recall | 10.18 (2.98) | 10.06 (2.68)
  Post-LIFUP Delayed Recall | 8.82 (3.43) | 8.47 (3.66)

2. Primary Outcome: State Trait Anxiety Inventory - State (STAIS)
Description: The "state" section of the State Trait Anxiety Inventory. This is a 20-question self-report assessment in which participants are asked about how they feel "right now, at this very moment" in order to assess current anxiety levels. Each item is scored on a scale of 1 to 4 points. The total assessment has a range of 20 to 80 points. Higher scores represent higher levels of anxiety.
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Population: All participants who completed this assessment before and after LIFUP at both the entorhinal cortex and the amygdala visits were included in analyses. One additional participant was removed due to presumed accidental reversal of the scale during the pre-LIFUP assessment, in which all of their responses were exactly flipped relative to their post-LIFUP responses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LIFUP to Entorhinal Cortex | LIFUP to Amygdala
Number analyzed (Participants) | 16 | 16
score on a scale
  STAIS Pre-LIFUP | 25.81 (6.67) | 30.69 (12.00)
  STAIS Post-LIFUP | 29.25 (10.64) | 30.63 (15.09)

3. Primary Outcome: Average Perfusion in Regions Of Interest
Description: Average perfusion in a given region of interest, as measured by arterial spin labeling. Percent change values calculated as ((Post LIFUP Perfusion - Pre LIFUP Perfusion)/Pre LIFUP Perfusion).
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Population: All participants who completed both pre and post-LIFUP arterial spin labeling scans at both visits
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | LIFUP to Entorhinal Cortex | LIFUP to Amygdala
Number analyzed (Participants) | 17 | 17
Percent
  Percent Change Perfusion in the Left Entorhinal Cortex | 15.75 (23) | 6.72 (34)
  Percent Change Perfusion in the Right Amygdala | 7.07 (35) | 19.52 (38)

4. Secondary Outcome: Emotional Reactivity Task
Description: An emotional reactivity and reappraisal task (ERT) using images from the International Picture Affective System (IAPS). Arousal ratings ranged from 1 (low arousal, "calm") to 9 (high arousal, "excited"). Valence ratings ranged from 1 (negative, "unhappy") to 9 (positive, "happy"). There were 3 instruction conditions: "WATCH", in which a participant was instructed to passively view a negatively-valenced image, "VIEW", in which they were instructed to passively view a neutral image, and "REAPPRAISE", in which participants were asked to change their emotional response to neutral in response to a negatively-valenced image by altering their cognitive construal of the image.
  The reported metric "reactivity" was taken from subtracting average responses to "VIEW" from average response to WATCH (i.e. WATCH - VIEW). Reappraisal metric is calculated as REAPPRAISE - WATCH
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Population: All participants who completed the IAPS ERT at all timepoints
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LIFUP to Entorhinal Cortex | LIFUP to Amygdala
Number analyzed (Participants) | 15 | 15
score on a scale
  Pre-LIFUP Reactivity - Arousal | 2.24 (2.78) | 2.20 (2.62)
  Post-LIFUP Reactivity - Arousal | 2.14 (2.98) | 3.02 (2.25)
  Pre-LIFUP Reappraisal - Arousal | -0.10 (0.55) | -0.18 (0.45)
  Post-LIFUP Reappraisal - Arousal | 0.22 (0.97) | -0.36 (0.94)
  Pre-LIFUP Reactivity - Valence | -3.06 (1.84) | -3.44 (1.31)
  Post-LIFUP Reactivity - Valence | -2.65 (3.14) | -3.21 (1.71)
  Pre-LIFUP Reappraisal - Valence | 0.54 (1.11) | 0.37 (0.87)
  Post-LIFUP Reappraisal - Valence | 0.07 (0.19) | 0.32 (0.83)

5. Secondary Outcome: Brief Visuospatial Memory Test
Description: Performance on the delayed recall (DR) portion of the Brief Visuospatial Memory Test (BVMT). Score is on a scale of 0-12, with higher scores indicating a better outcome. A score of 12 points represents full recall of all figures in their correct locations.
Time Frame: Pre-LIFUP and Post-LIFUP at Day 1 and Day 15
Population: All participants who completed the assessment at all time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LIFUP to Entorhinal Cortex | LIFUP to Amygdala
Number analyzed (Participants) | 16 | 16
score on a scale
  BVMT DR Pre-LIFUP | 9.63 (2.16) | 10.50 (1.41)
  BVMT DR Post-LIFUP | 8.56 (3.03) | 8.63 (2.83)

ADVERSE EVENTS:
Time Frame: Data was collected on Day 1 and Day 15
Arm/Group | Low Intensity Focused Ultrasound Pulsation to Amygdala | Low Intensity Focused Ultrasound Pulsation to Entorhinal Cortex
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/21 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Intensity Focused Ultrasound Pulsation to Amygdala (N=21) | Low Intensity Focused Ultrasound Pulsation to Entorhinal Cortex (N=21)
Emotional distress following sonication (Psychiatric disorders) | 1 (1) | 0 (0) — Visibly increased anxiety and general distress after sonication. Distress was transient and mostly resolved within a few hours. Unclear to what extent this resulted from treatment vs other possible etiologies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT03717922/Prot_SAP_003.pdf